CLINICAL TRIAL: NCT06490250
Title: Comparison of the Effects of Inspiratory Muscle Training and Baduanjin Exercises on Pulmonary Function, Exercise Capacity and Quality of Life in Patients With Hypertrophic Cardiomyopathy
Brief Title: Comparison of the Effects of Inspiratory Muscle Training and Baduanjin Exercises in Hypertrophic Cardiomyopathy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Muhammed Yurtseven, PhD Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC-FTR-MY-01
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hypertrophic Cardiomyopathy; Heart Diseases
Keywords: Exercise capacity; Pulmonary function; Quality of life
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Three groups with control group
Who Masked: Outcomes Assessor
Masking Description: Outcome assessments will be performed by an investigator who is blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inspiratory Muscle Training (IMT) Group (Experimental): The inspiratory muscle training group will participate in the respiratory exercise program with the IMT device.
  Interventions: Other: Inspiratory Muscle Training
- Baduanjin Exercise Group (Experimental): The Baduanjin group will participate in the Baduanjin exercise program, which includes 8 movements.
  Interventions: Other: Baduanjin Exercise
- Control Group (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Other: Inspiratory Muscle Training — The IMT group will use an inspiratory muscle training device twice a day, every day of the week, for 15 minutes. This training will continue for 8 weeks, with supervision once a week and unsupervised sessions on the other day
  Arms: Inspiratory Muscle Training (IMT) Group
Other: Baduanjin Exercise — The Baduanjin group will participate in a 50-minute exercise program, which includes a 10-minute warm-up, a 30-minute routine of eight separate movements, and a 10-minute cool-down. This will occur three times a week (twice in person and once online) for 8 weeks.
  Arms: Baduanjin Exercise Group

SUMMARY:
The study aims to compare the effects of inspiratory muscle training and Baduanjin exercises on pulmonary function, exercise capacity, and quality of life in patients with hypertrophic cardiomyopathy. By investigating these interventions, the investigators seek to introduce novel approaches that can enhance pulmonary function, exercise capacity, and overall quality of life for these patients.

In the study, which will involve three groups-the control group, the inspiratory muscle training (IMT) group, and the Baduanjin group-it was calculated that a total of 51 patients, with 17 in each group (n = 17), should be included.

The IMT group will use an inspiratory muscle training device twice a day, every day of the week, for 15 minutes. This training will continue for 8 weeks, with supervision once a week and unsupervised sessions on the other days.

The Baduanjin group will participate in a 50-minute exercise program, which includes a 10-minute warm-up, a 30-minute routine of eight separate movements, and a 10-minute cool-down. This will occur three times a week (twice in person and once online) for 8 weeks.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is characterized by a left ventricular wall thickness exceeding 15 millimeters (mm), as assessed by echocardiography and cardiac magnetic resonance imaging (MRI). It is a common genetic heart disease worldwide, known to cause left ventricular outflow tract obstruction, mitral regurgitation, diastolic dysfunction, myocardial ischemia, arrhythmias, and autonomic dysfunction (PubMed identification number (ID): 29655825, 28912181, 24998133, 30110588, 33229115).

Many patients with HCM are asymptomatic, and the condition is often identified incidentally during routine screening. Symptomatic patients may experience dyspnea on exertion, chest pain, syncope, or presyncope (PubMed ID:11886323). Even when left ventricular systolic function is preserved, patients frequently develop symptoms such as dyspnea and fatigue, leading to exercise intolerance in the majority (PubMed ID:10913477).

HCM is a heterogeneous disease with a varied clinical course. In addition to these symptoms, patients may also face decreased exercise capacity and reduced quality of life (PubMed ID:19253387, 9326995). Furthermore, despite the well-established cardiovascular and overall health benefits of regular physical activity, many patients with HCM exhibit a high prevalence of physical inactivity (PubMed ID: 23340032, 27547438).

Studies on inspiratory muscle training have demonstrated its benefits in improving respiratory function, respiratory muscle strength, quality of life, and exercise capacity across various patient groups including chronic obstructive pulmonary disease, cystic fibrosis, spinal cord injury, and heart failure. It also helps alleviate symptoms of dyspnea and fatigue (PubMed ID:32209709, 30827470, 32936904, 31429207, 31937553). Additionally, inspiratory muscle training has been shown to enhance physical activity levels in different patient cohorts (PubMed ID: 17534784).

Research indicates that Baduanjin exercises can serve as a complementary and alternative treatment for cardiovascular patients, improving clinical outcomes and reducing adverse cardiovascular events (PubMed ID:30059552). Furthermore, studies have highlighted their positive effects on quality of life and exercise capacity in diverse populations such as healthy individuals and those with conditions like heart failure, Parkinson's disease, osteoarthritis, and chronic fatigue syndrome, while also mitigating fatigue symptoms (PubMed ID: 36436262, 19051349, 27627031, 23001463, 18315512, 26083663, 25610473, 27938498).

Based on existing literature, the investigators believe that inspiratory muscle training and Baduanjin exercises could potentially benefit patients with HCM by alleviating associated symptoms. However, there is a notable scarcity of studies investigating different exercise modalities in HCM patients. To the investigators' knowledge, no studies have specifically examined the effects of inspiratory muscle training or Baduanjin exercises in this population.

The study aims to fill this gap by being the first to compare the impacts of inspiratory muscle training and Baduanjin exercises on pulmonary function, exercise capacity, and quality of life in patients with HCM. Through this research, the investigators seek to introduce new approaches that enhance pulmonary function, exercise capacity, and overall quality of life for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial thickness in any region of the left ventricle is 15 mm or more on echocardiography or cardiac MRI
* Clinically and hemodynamically stable (patients with NYHA Class I and II)
* Patients over 18 years of age
* Patients who provide informed consent

Exclusion Criteria:

* Acute decompensated heart failure
* Decreased ejection fraction (<40%)
* Unstable angina pectoris
* Significant coronary artery disease (CAD)
* Severe renal dysfunction (estimated glomerular filtration rate <30 mL/min/m²)
* Uncontrolled hypertension (despite medication)
* Severe valve disease (moderate-severe aortic stenosis, advanced mitral regurgitation)
* Severe neurological disorders causing autonomic dysfunction
* Cognitive impairment that prevents communication
* Recent fractures, osteoporosis, presence of tumors, pregnancy, or back and spine problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The Six-Minute Walk Test (6MWT) | Change from Baseline at 8 weeks
  Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society. Functional exercise capacity will be evaluated with the six-minute walk test. Patients will be walked in a 30-meter-long corridor for 6 minutes and the maximum walking distance will be measured. Before and after the test, heart rate, blood pressure and O2 saturation will be measured with pulse oximetry, and dyspnea and fatigue levels will be determined according to the Modified Borg scale.

SECONDARY OUTCOMES:
Pulmonary Function Tests (PFT) | Change from Baseline at 8 weeks
  Pulmonary function tests will be conducted using a spirometer, following the American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria.
Maximal Inspiratory Pressure (MIP) | Change from Baseline at 8 weeks
  Inspiratory muscle strength will be measured using a portable electronic oral pressure measurement device (MicroRPM; Micro Medical, UK). According to the recommendations of the American Thoracic Society and the European Respiratory Society, a maximum of five maneuvers will be performed, with 1-minute intervals between them. For maximum inspiratory pressure (MIP) measurement, patients will be seated and will first exhale maximally using a nose clip, then be asked to inhale maximally through a mouthpiece for at least 2 seconds. The results will be recorded in centimetres of water (cmH2O) and as a percentage of the expected value. Maneuvers will be considered satisfactory when a change of less than 10% is observed between three measurements, and the highest value will be recorded.
Nitric Oxide Levels | Change from Baseline at 8 weeks
  Nitric oxide levels' measurements will be performed with a fractional exhaled nitric oxide (FeNO) device.
Minnesota Living with Heart Failure Questionnaire | Change from Baseline at 8 weeks
  The Minnesota Living with Heart Failure Questionnaire will be used to assess the quality of life. This questionnaire evaluates how much heart failure has affected the patient's life over the past month (4 weeks). Patients circle a number from 0 to 5 next to each question to indicate the impact on their life, with 0 meaning no impact. The survey consists of 21 questions.
New York Heart Association (NYHA) Classification | Change from Baseline at 8 weeks
  The New York Heart Association (NYHA) Classification provides a simple way of classifying the extent of heart failure. It classifies patients in one of four categories based on their limitations during physical activity; the limitations/symptoms are in regards to normal breathing and varying degrees in shortness of breath and or angina pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rengin Demir, Prof, Study Director — Istanbul University-Cerrahpasa (IUC) Cardiology Institute; Veysel Oktay, Assoc Prof, Study Chair — Istanbul University-Cerrahpasa (IUC) Cardiology Institute
Locations (1):
- Istanbul University-Cerrahpasa (IUC) Cardiology Institute, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geske JB, Ommen SR, Gersh BJ. Hypertrophic Cardiomyopathy: Clinical Update. JACC Heart Fail. 2018 May;6(5):364-375. doi: 10.1016/j.jchf.2018.02.010. Epub 2018 Apr 11. PMID 29655825
- [Background] Marian AJ, Braunwald E. Hypertrophic Cardiomyopathy: Genetics, Pathogenesis, Clinical Manifestations, Diagnosis, and Therapy. Circ Res. 2017 Sep 15;121(7):749-770. doi: 10.1161/CIRCRESAHA.117.311059. PMID 28912181
- [Background] Maron BJ, Ommen SR, Semsarian C, Spirito P, Olivotto I, Maron MS. Hypertrophic cardiomyopathy: present and future, with translation into contemporary cardiovascular medicine. J Am Coll Cardiol. 2014 Jul 8;64(1):83-99. doi: 10.1016/j.jacc.2014.05.003. PMID 24998133
- [Background] Maron BJ. Clinical Course and Management of Hypertrophic Cardiomyopathy. N Engl J Med. 2018 Aug 16;379(7):655-668. doi: 10.1056/NEJMra1710575. No abstract available. PMID 30110588
- [Background] Ommen SR, Mital S, Burke MA, Day SM, Deswal A, Elliott P, Evanovich LL, Hung J, Joglar JA, Kantor P, Kimmelstiel C, Kittleson M, Link MS, Maron MS, Martinez MW, Miyake CY, Schaff HV, Semsarian C, Sorajja P. 2020 AHA/ACC Guideline for the Diagnosis and Treatment of Patients With Hypertrophic Cardiomyopathy: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2020 Dec 22;76(25):3022-3055. doi: 10.1016/j.jacc.2020.08.044. Epub 2020 Nov 20. PMID 33229115
- [Background] Maron BJ. Hypertrophic cardiomyopathy: a systematic review. JAMA. 2002 Mar 13;287(10):1308-20. doi: 10.1001/jama.287.10.1308. PMID 11886323
- [Background] Sharma S, Elliott P, Whyte G, Jones S, Mahon N, Whipp B, McKenna WJ. Utility of cardiopulmonary exercise in the assessment of clinical determinants of functional capacity in hypertrophic cardiomyopathy. Am J Cardiol. 2000 Jul 15;86(2):162-8. doi: 10.1016/s0002-9149(00)00854-7. PMID 10913477
- [Background] Christiaans I, van Langen IM, Birnie E, Bonsel GJ, Wilde AA, Smets EM. Quality of life and psychological distress in hypertrophic cardiomyopathy mutation carriers: a cross-sectional cohort study. Am J Med Genet A. 2009 Feb 15;149A(4):602-12. doi: 10.1002/ajmg.a.32710. PMID 19253387
- [Background] Cox S, O'Donoghue AC, McKenna WJ, Steptoe A. Health related quality of life and psychological wellbeing in patients with hypertrophic cardiomyopathy. Heart. 1997 Aug;78(2):182-7. doi: 10.1136/hrt.78.2.182. PMID 9326995
- [Background] Reineck E, Rolston B, Bragg-Gresham JL, Salberg L, Baty L, Kumar S, Wheeler MT, Ashley E, Saberi S, Day SM. Physical activity and other health behaviors in adults with hypertrophic cardiomyopathy. Am J Cardiol. 2013 Apr 1;111(7):1034-9. doi: 10.1016/j.amjcard.2012.12.018. Epub 2013 Jan 19. PMID 23340032
- [Background] Sweeting J, Ingles J, Timperio A, Patterson J, Ball K, Semsarian C. Physical activity in hypertrophic cardiomyopathy: prevalence of inactivity and perceived barriers. Open Heart. 2016 Jul 20;3(2):e000484. doi: 10.1136/openhrt-2016-000484. eCollection 2016. PMID 27547438
- [Background] Figueiredo RIN, Azambuja AM, Cureau FV, Sbruzzi G. Inspiratory Muscle Training in COPD. Respir Care. 2020 Aug;65(8):1189-1201. doi: 10.4187/respcare.07098. Epub 2020 Mar 24. PMID 32209709
- [Background] Zeren M, Cakir E, Gurses HN. Effects of inspiratory muscle training on postural stability, pulmonary function and functional capacity in children with cystic fibrosis: A randomised controlled trial. Respir Med. 2019 Mar;148:24-30. doi: 10.1016/j.rmed.2019.01.013. Epub 2019 Jan 28. PMID 30827470
- [Background] Azambuja ACM, de Oliveira LZ, Sbruzzi G. Inspiratory Muscle Training in Patients With Heart Failure: What Is New? Systematic Review and Meta-Analysis. Phys Ther. 2020 Dec 7;100(12):2099-2109. doi: 10.1093/ptj/pzaa171. PMID 32936904
- [Background] Hossein Pour AH, Gholami M, Saki M, Birjandi M. The effect of inspiratory muscle training on fatigue and dyspnea in patients with heart failure: A randomized, controlled trial. Jpn J Nurs Sci. 2020 Apr;17(2):e12290. doi: 10.1111/jjns.12290. Epub 2019 Aug 19. PMID 31429207
- [Background] Boswell-Ruys CL, Lewis CRH, Wijeysuriya NS, McBain RA, Lee BB, McKenzie DK, Gandevia SC, Butler JE. Impact of respiratory muscle training on respiratory muscle strength, respiratory function and quality of life in individuals with tetraplegia: a randomised clinical trial. Thorax. 2020 Mar;75(3):279-288. doi: 10.1136/thoraxjnl-2019-213917. Epub 2020 Jan 14. PMID 31937553
- [Background] Aznar-Lain S, Webster AL, Canete S, San Juan AF, Lopez Mojares LM, Perez M, Lucia A, Chicharro JL. Effects of inspiratory muscle training on exercise capacity and spontaneous physical activity in elderly subjects: a randomized controlled pilot trial. Int J Sports Med. 2007 Dec;28(12):1025-9. doi: 10.1055/s-2007-965077. Epub 2007 May 29. PMID 17534784
- [Background] Xiao X, Wang J, Gu Y, Cai Y, Ma L. Effect of community based practice of Baduanjin on self-efficacy of adults with cardiovascular diseases. PLoS One. 2018 Jul 30;13(7):e0200246. doi: 10.1371/journal.pone.0200246. eCollection 2018. PMID 30059552
- [Background] Yang WY, Xu Y, Ye L, Rong LJ, Feng J, Huang BL, Chien CW, Tung TH. Effects of Baduanjin exercise on quality-of-life and exercise capacity in patients with heart failure: A systematic review and meta-analysis. Complement Ther Clin Pract. 2023 Feb;50:101675. doi: 10.1016/j.ctcp.2022.101675. Epub 2022 Oct 28. PMID 36436262
- [Background] Hsu MC, Wang TS, Liu YP, Liu CF. Effects of Baduanjin exercise on oxidative stress and antioxidant status and improving quality of life among middle-aged women. Am J Chin Med. 2008;36(5):815-26. doi: 10.1142/S0192415X08006260. PMID 19051349
- [Background] Xiao C, Zhuang Y, Kang Y. Effect of Health Qigong Baduanjin on Fall Prevention in Individuals with Parkinson's Disease. J Am Geriatr Soc. 2016 Nov;64(11):e227-e228. doi: 10.1111/jgs.14438. Epub 2016 Sep 14. No abstract available. PMID 27627031
- [Background] An BC, Wang Y, Jiang X, Lu HS, Fang ZY, Wang Y, Dai KR. Effects of Baduanjin () exercise on knee osteoarthritis: a one-year study. Chin J Integr Med. 2013 Feb;19(2):143-8. doi: 10.1007/s11655-012-1211-y. Epub 2012 Sep 21. PMID 23001463
- [Background] An B, Dai K, Zhu Z, Wang Y, Hao Y, Tang T, Yan H. Baduanjin alleviates the symptoms of knee osteoarthritis. J Altern Complement Med. 2008 Mar;14(2):167-74. doi: 10.1089/acm.2007.0600. PMID 18315512
- [Background] Liao Y, Lin Y, Zhang C, Xue XL, Mao QX, Zhang Y, Dai JG, Wang TF. Intervention Effect of Baduanjin Exercise on the Fatigue State in People with Fatigue-Predominant Subhealth: A Cohort Study. J Altern Complement Med. 2015 Sep;21(9):554-62. doi: 10.1089/acm.2014.0395. Epub 2015 Jun 17. PMID 26083663
- [Background] Chan JS, Ho RT, Chung KF, Wang CW, Yao TJ, Ng SM, Chan CL. Qigong exercise alleviates fatigue, anxiety, and depressive symptoms, improves sleep quality, and shortens sleep latency in persons with chronic fatigue syndrome-like illness. Evid Based Complement Alternat Med. 2014;2014:106048. doi: 10.1155/2014/106048. Epub 2014 Dec 25. PMID 25610473
- [Background] Chan JS, Li A, Ng SM, Ho RT, Xu A, Yao TJ, Wang XM, So KF, Chan CL. Adiponectin Potentially Contributes to the Antidepressive Effects of Baduanjin Qigong Exercise in Women With Chronic Fatigue Syndrome-Like Illness. Cell Transplant. 2017 Mar 13;26(3):493-501. doi: 10.3727/096368916X694238. Epub 2016 Dec 7. PMID 27938498